CLINICAL TRIAL: NCT01136928
Title: Phase I Pharmacokinetic Interaction Study of Efavirenz and American Ginseng in Healthy Volunteers
Brief Title: Pharmacokinetic Interaction Study of Efavirenz and American Ginseng in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00038067; R01AT005526-01 (NIH)
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: Antiretroviral therapy; American ginseng; Efavirenz; Cytochrome P450 enzymes; Complementary and Alternative Medicine; Herbal; Pharmacikinetics; Healthy volunteers
MeSH Terms: interventions — Asian ginseng; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- American ginseng and efavirenz (Experimental): This is a sequential study. Healthy volunteers will receive efavirenz alone for 14 days followed by efavirenz plus American ginseng for an additional 14 days.
  Interventions: Drug: American ginseng

INTERVENTIONS:
Drug: American ginseng — Healthy volunteers will ge given efavirnez 600 mg daily monotherapy for 14 days followed by efavirenz 600 mg PLUS American ginseng 3000 mg daily for an additional 14 days.
  Other Names: Efavienz (Sustiva)

SUMMARY:
This is a 4-week sequential drug interaction study to measure the effects of American ginseng on efavirenz pharmacokinetics using steady-state 24-hour Area Under the Curve (AUC) and Cmax as the primary comparison measures in healthy male volunteers. Efavirenz Cmin, T1/2, tmax, and clearance will also be assessed as secondary outcome measures. This study is a phase I, prospective, within-subject, fixed-order, two-period, multiple dose, open label, drug interaction study, to determine the stead-state plasma pharmacokinetic profile of efavirenz before and after concurrent treatment with American ginseng. The investigators hypothesis is that concurrent oral administration of American ginseng for up to 14 days will not significantly alter the steady-state plasma pharmacokinetic of efavirenz.

DETAILED DESCRIPTION:
This study is supported by R01AT005526-01 grant awarded by National Center for Complementary and. Alternative Medicine (NCCAM) to evaluate the safety, efficacy, and mechanism of American ginseng in HIV-related fatigue. This is a 4-week sequential drug interaction study to measure the effects of American ginseng on efavirenz pharmacokinetics using steady-state 24-hour AUC and Cmax as the primary comparison measures in healthy male volunteers. Efavirenz Cmin, T1/2, tmax, and clearance will also be assessed as secondary outcome measures. This study is a phase I, prospective, within-subject, fixed-order, two-period, multiple dose, open label, drug interaction study, to determine the stead-state plasma pharmacokinetic profile of efavirenz before and after concurrent treatment with American ginseng. Therefore, this study will evaluate the effects of American ginseng on efavirenz plasma concentrations. Only efavirenz plasma concentrations will be measured in this study. American ginseng plasma concentrations will not be assessed in this study. Efavirenz plasma concentrations will be measured on study Days 14 and 28 (corresponding to weeks 2 and 4, respectively).

This is an important study because although American ginseng is a popular dietary supplement, the safety and efficacy of this agent in HIV-infected patients has not yet been established. A major concern regarding the safety of American ginseng in HIV-infected patients is the potential for herb-drug interactions that could alter the metabolism of antiretroviral drugs. Induction of drug metabolizing enzymes by dietary supplements such as American ginseng, could lead to a reduction in the therapeutic concentrations of these drugs and treatment failure. Inhibition of these drug metabolizing enzymes, on the other hand, could result in higher plasma concentrations of antiretroviral agents and potentially lead to increased toxicity.

Most antiretroviral drugs are metabolized by the cytochrome P450 (CYP450) isoenzyme CYP3A4. Our preliminary data suggest that American ginseng does not significantly affect CYP3A4 activity in vivo. A recent study has also reported that the American ginseng-mediated induction of Uridyl dipohsphate (UDP)-glucuronosyltransferase enzyme involved in the metabolism of the nucleoside reverse transcriptase inhibitors (NRTIs) zidovudine and abacavir, and the integrase inhibitor raltegravir, does not significantly alter zidoduvine pharmacokinetics. However, data are not available concerning the effect of American ginseng on other major CYP 450 isoforms involved in the metabolism of antiretroviral drugs. For instance, the non- nucleoside reverse transcriptase inhibitor (NNRTI) efavirenz is also metabolized by CYP2B6 and only to a lesser extent by the CYP3A4 isoform. Therefore, a potential drug interaction between American ginseng and this popular NNRTI must be excluded before this herb can be safely used in HIV-infected patients. This study will complete the work that has been currently done characterizing the effects of American ginseng on major drug metabolizing enzymes.

DURATION:

The total duration of this study is five weeks. Participants will receive study medications during the first four weeks of the study. On week 5 participants will complete their final post treatment safety study visit.

POPULATION AND SAMPLE SIZE:

Fifteen adult healthy male volunteers will be enrolled in this study.

REGIMEN:

Period 1 Days 0-14 Daily efavirenz monotherapy 600 mg orally Efavirenz pharmacokinetic sampling on Day 14

Period 2 Days 15-28 Daily efavirenz 600 mg orally PLUS American ginseng 3000 mg orally Efavirenz pharmacokinetic sampling on Day 28

Because efavirenz is a Category D drug with positive evidence of fetal risk, only male healthy volunteers will be enrolled in this study. Our hypothesis is that concurrent oral administration of American ginseng for up to 14 days will not significantly alter the steady-state plasma pharmacokinetic of efavirenz.

ELIGIBILITY:
Inclusion Criteria:

1. All enrollees will be healthy volunteers, ≥18 years of age with
2. Negative HIV-1 serology, documented by any licensed ELISA test kit
3. Ability and willingness to provide a signed informed consent and comply with study requirements
4. Males only because efavirenz has been reported to have teratogenic properties
5. Estimated creatinine clearance ≥50 mL/minute, as calculated by the Cockcroft-Gault method
6. Normal laboratory and physical examination, as judged by the Principal Investigator
7. Good peripheral venous access
8. Willingness and ability to take oral medications.

Exclusion Criteria:

1. Known or suspected hypersensitivity to American Ginseng (AG) or efavirenz
2. Taking any prescription, over-the-counter medication, or Complementary and alternative medicine (CAM) agents within 30 days of study enrolment
3. Evidence of active drug or alcohol abuse
4. Any other medical or psychological condition that might, in the opinion of the investigator, interfere with participation in the study or put subjects at undue risk
5. Hospitalization or therapy for serious illness within 30 days prior to study entry, as judged by the investigator
6. Participation in any investigational drug trials within 30 days prior to study entry that, in the opinion of the investigator, would preclude study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2011-03-14 (Actual); Study Completion 2011-03-14 (Actual)

PRIMARY OUTCOMES:
To compare efavirenz AUC0-24 and Cmax when dosed alone to steady-state efavirenz AUC0-24 and Cmax given concurrently with American ginseng. Efavirenz AUC0-24 with and without American ginseng | 14 days of efavirenz alone, followed by 14 days of concurrent administration of efavirenz and American ginseng
  Compare efavirenz AUC0-24 and Cmax when dosed alone at 600 mg daily, to steady-state efavirenz AUC0-24 and Cmax dosed at 600 mg daily and given concurrently with American ginseng 3000 mg daily.

SECONDARY OUTCOMES:
Efavirenz tmax with and without American ginseng | 14 days of efavirenz alone, followed by 14 days of concurrent administration of efavirenz and American ginseng
  To compare efavirenz tmax at steady-state when dosed alone as 600 mg daily, to steady-state efavirenz tmax dosed at 600 mg daily and given concurrently with American ginseng 3000 mg daily in HIV-seronegative healthy male volunteers.
Efavirenz Cmin with and without American ginseng | 14 days of efavirenz alone, followed by 14 days of concurrent administration of efavirenz and American ginseng
  To compare efavirenz Cmin at steady-state when dosed alone as 600 mg daily, to steady-state efavirenz Cmin dosed at 600 mg daily and given concurrently with American ginseng 3000 mg daily in HIV-seronegative healthy male volunteers.
Efavirenz Clearance with and without American ginseng | 14 days of efavirenz alone, followed by 14 days of concurrent administration of efavirenz and American ginseng
  To compare efavirenz Clearance at steady-state when dosed alone as 600 mg daily, to steady-state efavirenz Clearance dosed at 600 mg daily and given concurrently with American ginseng 3000 mg daily in HIV-seronegative healthy male volunteers
Efavirenz T1/2 with and without American ginseng | 14 days of efavirenz alone, followed by 14 days of concurrent administration of efavirenz and American ginseng
  To compare efavirenz T1/2 at steady-state when dosed alone as 600 mg daily, to steady-state efavirenz T1/2 dosed at 600 mg daily and given concurrently with American ginseng 3000 mg daily in HIV-seronegative healthy male volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Andrade, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States